CLINICAL TRIAL: NCT01623882
Title: Clinical Evaluation of the Combined Use of Apligraf® and the SNaP® Negative Pressure Wound Therapy System for Treatment of Non-responding Venous Stasis and Diabetic Lower Extremity Ulcers
Brief Title: Clinical Evaluation of the Combined Use of Apligraf® and the SNaP® Pressure Wound Therapy System
Acronym: OG/SNaP
Status: Withdrawn | Type: Observational
Why Stopped: The study was terminated by Spiracur (original sponsor). Efforts were made to contact the PI/study team members, but were unsuccessful.
Sponsor: KCI USA, Inc (Industry)
Collaborators: Organogenesis (Industry); 3M (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Other Study IDs: 041311
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes Mellitus; Wounds; Ulcers
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries; Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of the concurrent use of Apligraf® and the SNaP® Wound Care System for the treatment of diabetic and venous stasis lower extremity ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Wound < 10 cm in greatest diameter
* Wound age > 4 weeks and patient shows < 50% wound area healing after 4 weeks of treatment
* Patient > 18 years of age
* Patient is willing and able to sign consent
* Patient is willing and able to complete study visits and comply with study dressing protocols

Exclusion Criteria:

* Wound size reduction of > 50% in last 4 weeks of treatment
* Patients with active wound infections, including cellulitis and osteomyelitis
* Patients with wounds not able to have eschar debrided
* ABI < 0.65 or SPP < 30mmHg
* Patients with wounds in anatomic areas which preclude achieving an airtight seal for NPWT
* Ulcers due to inflammatory conditions such as rheumatoid arthritis, lupus, scleroderma, vasculitis, calciphylaxis, etc.
* Patients with allergy to or intolerance of any of the wound dressing materials expected to be used during the trial.
* Pregnant patients
* Patients unable to tolerate NPWT
* Patients with dialysis dependent ESRD
* Index ulcer is on the plantar surface of the foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower extremity venous and diabetic ulcers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of wounds closed | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schubart, MD, PhD, Principal Investigator — O'Connor Hospital